CLINICAL TRIAL: NCT06698900
Title: Generating Evidence Study for Systemic Lupus Erythematosus Using Different Types of Methodologies
Brief Title: This Project Aims to Understand the Needs of Rheumatologists and Other Specialties in the Care of Patients With SLE
Acronym: LESBRA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00089
Record Dates: First submitted 2024-10-21; First posted 2024-11-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Rheumatologists; Arthritis; Spondylitis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis; Spondylitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project will be conducted in four distinct stages. Firstly, evidence synthesis will be carried out to gather and analyze available data on the topic. Following this, a discussion among physicians will be facilitated to understand the knowledge gaps among rheumatologists and other specialists regarding SLE. Subsequently, consensus will be sought among a select group of rheumatologists on various aspects related to patient care, unmet medical needs, and implementation of new technologies. Finally, the findings and conclusions from these stages will be used to inform the development and publication of scientific papers.

DETAILED DESCRIPTION:
This study has as geral objective understanding the currently unmet development needs of rheumatologists and other specialists involved in the care of patients with SLE, from a comparative perspective with other rheumatic diseases. The goal is to increase the engagement of these professionals in the discussion and management of patients and sécific objectives, compare the currently available evidence on SLE and three other rheumatic diseases (rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis); Promote discussions to understand the knowledge development needs of rheumatologists regarding SLE; Generate a consensus on the equity of rheumatic diseases in relation to public policies, guidelines, registries, patient association mobilization, patient journey, time to diagnosis, and available medications with access to treatment and, Promote awareness and knowledge through scientific publications about SLE.

ELIGIBILITY:
Inclusion Criteria:

- All the patients with SLE registered in DataSUS, in the outpatient system (SIA) and in the Hospital System (SIH) from 2019 to 2022

Exclusion Criteria:

* Not applicable

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All population data identified in the literature review and desk research; analysis of the National Health Database in Brazil (DataSUS)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-11-29 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Understand the difficulties faced by patients with SLE and identify gaps in diagnosis and treatment | through study completion, an average of 3 months
  Prepare an evidence synthesis using available data, discuss the topic with medical experts to understand knowledge gaps among rheumatologists and other professionals regarding SLE, and build consensus among a group on various aspects related to patient care, unmet medical needs, and implementation of new technologies

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Monticielo OA, Seguro LPC, de Ataide Mariz H, Daher Macedo M, Therumi Assao V, Lima J, Volpi E Silva N, Dos Reis-Neto ET. Current landscape of immune-mediated inflammatory rheumatic diseases in Brazil's public and private systems: retrospective cohort study. BMJ Open. 2025 Nov 23;15(11):e104870. doi: 10.1136/bmjopen-2025-104870. PMID 41285502
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3461R00089&attachmentIdentifier=bb781b4f-1f4d-40eb-9e2d-d8a13a5c5c42&fileName=Clinical_Study_Report_CSR_Synopsis_LESBRA.pdf&versionIdentifier=